CLINICAL TRIAL: NCT01623765
Title: Diagnosis and Staging of Lung Cancer Using Minimally Invasive Technique With Ultrasound Guidance
Brief Title: Lung Cancer Diagnosis and Staging Using Ultrasound Guidance
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/458/B
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer
Keywords: Endobronchial ultrasound, lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To collect data of all patients who have undergone Endobronchial ultrasound for diagnosis or staging of suspected lung cancer

DETAILED DESCRIPTION:
Introduction: Endobronchial Ultrasound (EBUS) is a procedure that is performed via flexible bronchoscopy under moderate sedation for visualization of lymph nodes in the chest and biopsy under real-time guidance for the staging of lung cancer or evaluation of enlarged lymph nodes. In addition, lung lesions or masses can be visualized and biopsied in the same sitting. The use of EBUS has enhanced the safety and diagnostic yield of flexible bronchoscopy.

Aim: The data of patients with suspected lung cancer or undiagnosed lymph node enlargement in whom bronchoscopy with EBUS guidance is clinically indicated will be collected prospectively.

Results from EBUS are considered positive if a specific diagnosis is obtained ( eg malignancy) or if lymphocytes are present in the lymph node biopsy, indicating accurate sampling of lymph node. In patients with non-diagnostic EBUS, the results from other procedures will be compared for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone endobronchial ultrasound

Exclusion Criteria: None

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore